CLINICAL TRIAL: NCT07280884
Title: Effect of Hemiparesis Side on Physiotherapy Outcomes Using the Luna EMG in Post-Ischemic Stroke Patients
Brief Title: Effect of Luna EMG Robotic Therapy on Physiotherapy Outcomes in Post-Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Collaborators: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 153/MN/IRK/2022
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke; Hemiparesis; Gait Disorders
Keywords: Physiotherapy; Robotic rehabilitation; Luna EMG
MeSH Terms: conditions — Ischemic Stroke; Paresis; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Luna EMG) (Experimental): 20 minutes of training using Luna EMG (reactive EMG-controlled knee extensions/flexions, CPM exercises, EMG biofeedback isometric exercises), 3 times a week for 4 weeks. PLUS Standard Rehabilitation.
  Interventions: Device: Luna EMG Robotic Training; Procedure: Conventional Physiotherapy
- Control Group (Standard Therapy) (Active Comparator): Active resistance exercises for 20 minutes (mirroring the time of the experimental group), 3 times a week, alongside the standard rehabilitation program (2 hours/day total)
  Interventions: Procedure: Conventional Physiotherapy

INTERVENTIONS:
Device: Luna EMG Robotic Training — Therapy utilizing the Luna EMG robot (EgzoTech, Gliwice, Poland) performed 3 times a week for 20 minutes over 4 weeks. The training utilizes reactive electromyography to capture muscle signals and facilitate movement. The session protocol includes:
  Reactive EMG Trigger & Hold (Knee Extension) - 5 mins. Continuous Passive Motion (CPM) - 1 min. Reactive EMG Trigger & Hold (Knee Flexion) - 5 mins. Continuous Passive Motion (CPM) - 1 min. EMG Biofeedback (Isometric exercises for knee extensors and flexors) - 8 mins.
  Arms: Experimental Group (Luna EMG)
Procedure: Conventional Physiotherapy — Standard neurological rehabilitation program conducted 2 hours daily, 6 times a week for 4 weeks. The program includes trunk stabilization, gait re-education (PNF method), manual dexterity exercises, and balance/coordination training. For the Control Group: During the time corresponding to robotic training, patients performed active resistance exercises for the lower limb for 20 minutes.

SUMMARY:
The study evaluates the effectiveness of the Luna EMG robotic system in the rehabilitation of patients after ischemic stroke. The main objective is to assess the impact of robotic-assisted training on gait speed, balance, and bioelectrical activity of the thigh muscles (rectus femoris and biceps femoris). The study also analyzes whether the side of hemiparesis (left vs. right) influences the outcomes of physiotherapy. Participants are randomly assigned to either an experimental group receiving robotic therapy combined with standard rehabilitation or a control group receiving standard rehabilitation alone.

DETAILED DESCRIPTION:
This prospective, randomized clinical trial aims to determine the efficacy of Luna EMG-assisted training in post-stroke motor recovery. The study involves 62 patients aged 65-86 years recovering from ischemic stroke (4-15 weeks post-stroke).

Participants are randomized into two groups:

Experimental Group: Patients undergo a 4-week rehabilitation program consisting of standard physiotherapy (2 hours/day, 6 days/week) combined with robotic training using the Luna EMG device (20 minutes, 3 days/week). The robotic protocol includes reactive EMG-triggered exercises, continuous passive motion (CPM), and EMG biofeedback isometric exercises.

Control Group: Patients undergo the same standard physiotherapy program (2 hours/day, 6 days/week) but perform active resistance exercises instead of robotic training during the equivalent time slots.

The primary outcome measures include balance assessment (Timed Up and Go, Berg Balance Scale, Trunk Impairment Scale, Postural Assessment Scale for Stroke Patients) and gait speed (10-Meter Walk Test). Secondary outcomes involve the analysis of surface electromyography (sEMG) signals from the paretic lower limb muscles to evaluate changes in bioelectrical activity. The study specifically investigates comparative outcomes between patients with left-sided versus right-sided hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary ischemic stroke
* Time from stroke: 4 to 15 weeks
* Age between 65 and 86 years
* Limited or impaired lower limb function
* Ability to walk 10 meters independently or with orthopedic assistance
* Muscle strength of at least -3 on the modified Medical Research Council (MRC) scale
* Cognitive function sufficient to understand instructions and participate in the study
* Stable clinical status
* Provided written informed consent

Exclusion Criteria:

* Hemorrhagic stroke or stroke in the posterior cerebral circulation
* Lower limb spasticity greater than 1+ on the modified Ashworth Scale (MAS)
* Functional limitations preventing the completion of selected tests
* Recent orthopedic injuries affecting balance
* Prior lower limb surgery
* Sensory aphasia
* Coexisting neurological disorders (e.g., Parkinson's disease, Huntington's disease)
* Lack of patient cooperation or refusal to consent

Ages: 65 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Static and Dynamic Balance (Berg Balance Scale - BBS) | Baseline and at 4 weeks (post-intervention)
  The BBS is a 14-item objective measure that assesses static balance and fall risk in adult populations. Tasks include sitting to standing, standing unsupported, reaching, turning, etc. The score ranges from 0 to 56, where higher scores indicate better balance.
Change in Functional Mobility and Balance (Timed Up and Go Test - TUG) | Baseline and at 4 weeks (post-intervention)
  The TUG test assesses mobility, balance, walking ability, and fall risk. The patient stands up from a chair, walks 3 meters, turns around, walks back, and sits down. The time taken to complete the task is measured in seconds. Lower time indicates better functional mobility.
Change in Trunk Control (Trunk Impairment Scale - TIS) | Baseline and at 4 weeks (post-intervention)
  The TIS evaluates motor impairment of the trunk after stroke. It assesses static sitting balance, dynamic sitting balance, and coordination. Higher scores indicate better trunk control and stability.
Change in Postural Control (Postural Assessment Scale for Stroke Patients - PASS) | Baseline and at 4 weeks (post-intervention)
  The PASS assesses postural control in patients after stroke. It measures the ability to maintain and change lying, sitting, and standing postures. Higher scores indicate better postural performance.
Change in Gait Speed (10-Meter Walk Test - 10MWT) | Baseline and at 4 weeks (post-intervention)
  Assesses walking speed over a short distance. The patient walks 10 meters, and the time is measured for the intermediate 6 meters to allow for acceleration and deceleration. The result is calculated in meters per second (m/s). Higher speed indicates better gait performance.

SECONDARY OUTCOMES:
Change in Bioelectrical Activity of the Rectus Femoris Muscle | Baseline and at 4 weeks (post-intervention)
  Measured using surface electromyography (sEMG) with the Luna EMG system. The mean amplitude of the sEMG signal is recorded during active knee extension of the paretic limb to assess muscle activation. Measured in microvolts (µV).
Change in Bioelectrical Activity of the Biceps Femoris Muscle | Baseline and at 4 weeks (post-intervention)
  Measured using surface electromyography (sEMG) with the Luna EMG system. The mean amplitude of the sEMG signal is recorded during active knee flexion of the paretic limb to assess muscle activation. Measured in microvolts (µV).

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Sihinkiewicz, PhD, Principal Investigator — Andrzej Frycz Modrzewski Krakow University
Locations (1):
- Non-Public Health Care Center "Rehstab" (NZOZ "RehStab"), Limanowa, Poland